CLINICAL TRIAL: NCT00285857
Title: A Phase 2 Trial of Lovastatin for Modification of Abnormal Breast Duct Cytology and Risk-Associated Biomarkers in Women at High Inherited Risk of Breast Cancer
Brief Title: Phase 2 Study of Lovastatin as Breast Cancer Chemoprevention
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, James Ford, Associate Professor of Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-13732; BRSNSTU0010 (Other: OnCore); 95505 (Other: Stanford University Alternate IRB Approval Number)
Record Dates: First submitted 2006-01-31; First posted 2006-02-02 (Estimated); Results first posted 2017-03-09 (Actual); Last update posted 2017-03-09 (Actual); Status verified 2017-01

CONDITIONS: Breast Cancer
Keywords: duct cytology
MeSH Terms: conditions — Breast Neoplasms | interventions — Lovastatin; lovastatin-niacin combination; Niacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lovastatin 80 mg/day (Experimental): Lovastatin 80 mg/day as 40 mg orally twice daily, for 6 months.
  Interventions: Drug: Lovastatin

INTERVENTIONS:
Drug: Lovastatin — Lovastatin 80 mg/day as 40 mg orally twice daily.
  Lovastatin is approved by FDA as a cholesterol-lowering agent.
  Other Names: Mevacor; Advicor (as a combination with niacin); Altocor; Altoprev; Statosan (Atos Pharma)

SUMMARY:
The study evaluates if a 6-month course of oral lovastatin at 80 mg/day would decrease abnormal breast duct cytology in women with a high inherited breast cancer risk.

DETAILED DESCRIPTION:
The study evaluates if a 6-month course of oral lovastatin at 80 mg/day (as 40 mg twice-a-day) would decrease abnormal breast duct cytology in women with a high inherited breast cancer risk. Breast duct cytology was assessed as hyperplasia or hyperplasia with atypia, as measured by random periareolar fine needle aspiration (rpFNA), of breast duct cells.

A stratified analysis of this objective will be performed according to BRCA mutation status (absence or presence of an inherited deleterious BRCA1 or BRCA2 mutation).

Additional objectives of the study are to:

* Assess change in mammographic density, which is known to associate with breast cancer risk, before and after treatment with lovastatin
* Asess incidence of breast cancers and new high-risk breast lesions, including atypical hyperplasia, ductal or lobular carcinoma in situ, or radial scar.
* Assess change in other breast cancer risk-associated biomarkers in rpFNA specimens, including:

  * Ki-67 (a marker of cell proliferation)
  * Estrogen receptor (ER)
  * Progesterone receptor (PR)
  * HER/2-neu over-expression
  * Susceptibility to DNA damage

ELIGIBILITY:
INCLUSION CRITERIA

* Female
* Increased inherited risk of breast cancer, as defined by:

  * Known deleterious mutation in BRCA1, BRCA2, or other high-risk mutation
  * Family history conveying at least a 2-fold increase in breast cancer risk
* ECOG performance status 0
* Normal organ and marrow function, including complete blood count and comprehensive metabolic panel within normal institutional limits
* Subject agreement to limit alcoholic beverage consumption to three alcoholic drinks per week.

EXCLUSION CRITERIA

* Prior history of invasive breast cancer less than 2 years previously (EXCEPTION: stage III or lower breast cancer > 2 years ago)
* Current or history of other cancers (EXCEPTION: non-melanoma skin cancer, or stage III or cancer without evidence of recurrence for 5 years
* Initial mammogram, breast MRI, or clinical breast examination prompts recommendation for biopsy by study investigators.
* Evidence of malignant cytology on initial rpFNA.
* Use of other investigational agents.
* Use of tamoxifen or selective estrogen response modifiers (SERMS), including raloxifene, within the last 2 years.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to lovastatin.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection; symptomatic congestive heart failure; unstable angina pectoris; cardiac arrhythmia; or psychiatric illness/social situations that would limit compliance with study requirements.
* Currently receiving lovastatin and cyclosporine, gemfibrozil, erythromycin, fibrates or niacin, (unless discontinued for study participation)
* No evidence of active liver disease, nor elevation of serum transaminases (prior history of liver disease, if not currently active, is not an exclusion)
* No evidence of myopathy or myositis, including symptoms of generalized muscle aches or weakness, muscle tenderness, or elevation in creatine phosphokinase.
* Lactating (breastfeeding)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-11; Primary Completion 2010-05 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Ford, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University Cancer Center, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vinayak S, Schwartz EJ, Jensen K, Lipson J, Alli E, McPherson L, Fernandez AM, Sharma VB, Staton A, Mills MA, Schackmann EA, Telli ML, Kardashian A, Ford JM, Kurian AW. A clinical trial of lovastatin for modification of biomarkers associated with breast cancer risk. Breast Cancer Res Treat. 2013 Nov;142(2):389-98. doi: 10.1007/s10549-013-2739-z. Epub 2013 Oct 29. PMID 24166281

RESULTS

PARTICIPANT FLOW:
Groups:
- Lovastatin 80 mg/Day: Lovastatin 80 mg/day given as 40 mg orally twice per day
Period: Overall Study
Arm/Group | Lovastatin 80 mg/Day
Started | 30
Completed | 26
Not Completed | 4
Not completed — Withdrawal by Subject | 2
Not completed — Inadequate initial breast cytology | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- Lovastatin: Lovastatin: 80 mg; 40 mg orally twice per day
Arm/Group | Lovastatin
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 45 [25 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Change in the Incidence of Abnormal Breast Duct Cytology After Treatment With Lovastatin 80 mg/Day
Description: Assessed on that basis of pre- and post-treatment evaluation with RPFNA (random periareolar fine needle aspiration). All subjects received a prescription for lovastatin 80 mg/day, to be taken as 40 mg twice-a-day.
  Cytology was qualitatively and quantitatively, using the Masood semiquantitative scale to assign a number to each specimen, with higher numbers indicating increasing degrees of abnormality, as follows:
  06-10 Non-proliferative breast disease (NPBD)
  11-14 Proliferative breast disease without atypia (PBD-A)
  15-18 Proliferative breast disease with atypia (PBD+A)
  19-24 Carcinoma in situ and invasive cancer (CIS/IC)
  If no cells could be obtained after multiple RPFNA attempts, the classification was acellular.
  Change from NPBD to PBD-A was considered Unfavorable.
  Change from NPBD to Acellular was considered Equivocal.
  Change from PBD-A to NPBD was considered Favorable.
Time Frame: 6 months
Population: Participants either at least one of the following:
  * Deleterious germline mutation in BRCA1, BRCA2, CDH1, or TP53
  * Lifetime breast cancer risk of breast cancer of 20 % as estimated by the Claus model
  * Personal history of estrogen receptor andprogesterone receptor-negative breast cancer.
Measure: Number; unit: participants
Groups:
- Baseline Non-proliferative Breast Disease (NPBD): Those subjects whose pre-treatment evaluation by RPFNA (random periareolar fine needle aspiration) returned a diagnosis of non-proliferative breast disease
- Baseline Proliferative Breast Disease Without Atypia (PBD-A): Those subjects whose pre-treatment evaluation by RPFNA (random periareolar fine needle aspiration) returned a diagnosis of proliferative breast disease without atypia
- Baseline Proliferative Breast Disease With Atypia (PBD+A): Those subjects whose pre-treatment evaluation by RPFNA (random periareolar fine needle aspiration) returned a diagnosis of proliferative breast disease with atypia
- Baseline Carcinoma in Situ or Invasive Cancer (CIS/IC): Those subjects whose pre-treatment evaluation by RPFNA (random periareolar fine needle aspiration) returned a diagnosis of carcinoma in situ or invasive cancer
- Baseline Biopsy Acellular: Those subjects whose pre-treatment evaluation by RPFNA (random periareolar fine needle aspiration) generated a sample that was acellular
Arm/Group | Baseline Non-proliferative Breast Disease (NPBD) | Baseline Proliferative Breast Disease Without Atypia (PBD-A) | Baseline Proliferative Breast Disease With Atypia (PBD+A) | Baseline Carcinoma in Situ or Invasive Cancer (CIS/IC) | Baseline Biopsy Acellular
Number analyzed (Participants) | 13 | 12 | 0 | 0 | 1
participants
  Post-treatment NPBD | 8 | 5 |  |  | 1
  Post-treatment PBD-A | 2 | 7 |  |  | 0
  Post-treatment PBD+A | 0 | 0 |  |  | 0
  Post-treatment CIS/IC | 0 | 0 |  |  | 0
  Post-treatment biopsy acellular | 3 | 0 |  |  | 0

2. Secondary Outcome: Change in Mammographic Density Before and After Treatment With Lovastatin 80 mg/Day
Description: Bilateral mammography was performed at study entry (before lovastatin therapy) and at study conclusion (after lovastatin therapy) . Mammograms were assessed for a decline in mean breast density, using the American College of Radiology Breast Imaging Reporting and Data System (BI-RAD) composition system for mammographic density assessment.
  Category 0 Need additional imaging evaluation
  1. Negative
  2. Benign
  3. Probably benign
  4. Suspicious abnormality
  5. Highly suggestive of malignancy
  6. Known biopsy-proven malignancy
Time Frame: 6 months
Population: Outcome reported as the change in mean mammographic density with standard deviation (SD) of the post-treatment measurements.
Measure: Mean (Standard Deviation); unit: BI-RADS
Arm/Group | Lovastatin 80 mg/Day
Number analyzed (Participants) | 30
BI-RADS | -0.10 (1.08)

3. Secondary Outcome: Change in Total Cholesterol After Treatment With Lovastatin 80 mg/Day
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Lovastatin 80 mg/Day
Number analyzed (Participants) | 25
mg/dL | -8 (45.7)

4. Secondary Outcome: Change in Low Density Lipoprotein (LDL) After Treatment With Lovastatin 80 mg/Day
Time Frame: 6 months
Population: Change in mean of LDL level, with standard deviation of the values at
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Lovastatin 80 mg/Day
Number analyzed (Participants) | 26
mg/dL | -6 (32.1)

ADVERSE EVENTS:
Arm/Group | Lovastatin
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 3/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lovastatin (N=30)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No